CLINICAL TRIAL: NCT02272647
Title: Progesterone Amplifies Estrogen-stimulated Growth Hormone Secretion in Older Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johannes D. Veldhuis, Professor, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-002829
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Normal Healthy Volunteers
MeSH Terms: interventions — Progesterone; Ghrelin; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IM Plac - Oral Plac - Ghrelin (Experimental): Day 1: IM Saline Placebo (0.25 ml) Day 10: IM Saline Placebo (0.5 ml) and Oral Placebo 3x/day Day 23: IV push of ghrelin (0.3 ug/kg) + Placebo (for 10 days)
  Interventions: Drug: IM Saline Placebo (0.25 ml); Drug: IM Saline Placebo (0.5 ml); Drug: Oral Placebo; Drug: Ghrelin (0.3 ug/kg)
- IM Plac - Oral Prog - Ghrelin (Experimental): Day 1: IM Saline Placebo (0.25 ml) Day 10: IM Saline Placebo (0.5 ml) and Oral Micronized Progesterone 3x/day Day 23: IV push of ghrelin (0.3 ug/kg) + Placebo (for 10 days)
  Interventions: Drug: IM Saline Placebo (0.25 ml); Drug: IM Saline Placebo (0.5 ml); Drug: Oral Micronized Progesterone; Drug: Ghrelin (0.3 ug/kg); Drug: Oral Placebo
- IM E2 - Oral Plac - Ghrelin (Experimental): Day 1: IM Estradiol (2.5 mg) Day 10: IM Estradiol (5.0 mg) and Oral Placebo 3x/day Day 23: IV push of ghrelin (0.3 ug/kg) + Medroxyprogesterone (5 mg - for 10 days)
  Interventions: Drug: IM Estradiol valerate (2.5 mg); Drug: IM Estradiol valerate (5.0 mg); Drug: Oral Placebo; Drug: Ghrelin (0.3 ug/kg); Drug: Medroxyprogesterone - Acetate
- IM E2 - Oral Prog - Ghrelin (Experimental): Day 1: IM Estradiol (2.5 mg) Day 10: IM Estradiol (5.0 mg) and Oral Micronized Progesterone 3x/day Day 23: IV push of ghrelin (0.3 ug/kg) + Placebo (for 10 days)
  Interventions: Drug: IM Estradiol valerate (2.5 mg); Drug: IM Estradiol valerate (5.0 mg); Drug: Oral Micronized Progesterone; Drug: Ghrelin (0.3 ug/kg); Drug: Oral Placebo

INTERVENTIONS:
Drug: IM Saline Placebo (0.25 ml)
  Arms: IM Plac - Oral Plac - Ghrelin; IM Plac - Oral Prog - Ghrelin
Drug: IM Estradiol valerate (2.5 mg)
  Arms: IM E2 - Oral Plac - Ghrelin; IM E2 - Oral Prog - Ghrelin
Drug: IM Saline Placebo (0.5 ml)
  Arms: IM Plac - Oral Plac - Ghrelin; IM Plac - Oral Prog - Ghrelin
Drug: IM Estradiol valerate (5.0 mg)
  Arms: IM E2 - Oral Plac - Ghrelin; IM E2 - Oral Prog - Ghrelin
Drug: Oral Micronized Progesterone
  Arms: IM E2 - Oral Prog - Ghrelin; IM Plac - Oral Prog - Ghrelin
Drug: Oral Placebo
  Arms: IM E2 - Oral Plac - Ghrelin; IM Plac - Oral Plac - Ghrelin
Drug: Ghrelin (0.3 ug/kg)
Drug: Medroxyprogesterone - Acetate
  Arms: IM E2 - Oral Plac - Ghrelin
Drug: Oral Placebo — (in lieu of Medroxyprogesterone)
  Arms: IM E2 - Oral Prog - Ghrelin; IM Plac - Oral Plac - Ghrelin; IM Plac - Oral Prog - Ghrelin

SUMMARY:
Progesterone amplifies estrogen-stimulated Growth Hormone (GH) secretion in postmenopausal women. Preliminary data are sought to estimate statistical power for more detailed studies of this hypothesis.

DETAILED DESCRIPTION:
The systemic availability and orderly secretion patterns of GH and sex steroids decline in healthy aging men and women. The combined changes have substantial clinical implications to aging-related physical frailty, diminished aerobic capacity, sarcopenia, osteopenia, visceral adiposity, glucose intolerance, and reduced psychosocial wellbeing. Whereas androgen is considered the main trophic (anabolic) sex steroid, recent data demonstrate that certain tissues respond principally to GH and testosterone-derived estradiol, Estrogen (E2) (e.g. bone, brain, liver and pituitary). In principle, frailty may thus be associated with dual GH and sex-steroid deficiencies. Additionally, young, but not older healthy women secrete significant amounts of progesterone for approximately 14 days during the luteal phase of every menstrual cycle. When GH levels rise nearly two fold, the investigators hypothesize that progesterone potentiates the GH response to E2. This hypothesis arises from scattered indirect studies often using synthetic progestins with partial androgen agonism, instead of progesterone per se.

Because there is no basis for estimating statistical power for this novel paradigm, 40 women, 10 each in 4 groups, will be studied. The pilot data will be used to calculate statistical power for a definitive R01-based investigation of gender-specific distinctions in estrogen-regulated pituitary-hormone secretion.

ELIGIBILITY:
Inclusion Criteria:

* women ages 50 to 80
* postmenopausal as defined by: any combination of the following

  * Hormonally postmenopausal for 1 year
  * Lh greater than 15 IU/L, FSH greater than 30 IU/L
  * Total hysterectomy with oophorectomy greater than one year
  * Hysterectomy with ovaries preserved with hormone levels: Lh > 15 IU/L, FSH > 30 IU/L
* Following laboratory results with normal range, unless PI approves out of range values.
* BMI 18 to 35

Exclusion Criteria:

* structural hypothalamo-pituitary-gonadal disease
* endocrinopathy (diseases involving the following organs pituitary, thyroid, adrenals, ovaries, testes and pancreas), other than primary thyroid failure receiving replacement
* recent (within 2 weeks) estrogen, progestin, anabolic steroid or glucocorticoid use
* clinically significant ECG abnormality as determined by study team physicians
* obstructive uropathy
* history of a stroke
* history of MI or angina
* acute or chronic systemic disease
* recent transmeridian travel (traversing more than 3 time zones within 7 days of admission)
* current night shift work
* concurrent use of neuropsychiatric medications
* alcohol or drug abuse, current and within 2 years
* history of depression, psychosis, or mania
* weight gain or loss (2 kg or more in 3 weeks)
* BMI > 35 kg/m2
* anemia, hemoglobin less than 12.5 g/dl
* abnormal hepatorenal function, creatinine outside normal range, ALT greater than two times normal range
* biochemical and chemistry lab results out of physician acceptable range
* history of deep-vein thrombophlebitis
* history of Congestive Heart Failure, cardiac arrhythmias, and medications used to treat cardiac arrhythmias
* known allergy to estradiol valerate, castor oil or sesame oil
* history of smoking within the last 2 years
* untreated gall bladder disease
* lack of voluntary, written informed consent
* history of carcinoma excluding localized basal cell or squamous cell, including women with known, suspected or history of breast cancer
* not clinically postmenopausal
* women with allergies to nuts will not be enrolled in the study.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Logarithm of the ratio of the normalized growth hormone secretion rate over the first 10 hr. | The subject will be followed on average for a month. Growth hormone measurements will occur on Day 23 after initiation of study drug administration
  Subjects will be given IM placebo/estradiol on Day 1. 10 days later they will receive IM placebo/estradiol again, then start progesterone/placebo capsules for 14 days. On Day 23, subjects will undergo a 12-h overnight (2200 - 1000h) fasting, 10-min blood sampling. The primary comparison parameter is the logarithm of the ratio of the normalized growth hormone secretion rate over the first 10 hr.

SECONDARY OUTCOMES:
Growth hormone secretion post ghrelin injection | The subject will be followed on average for a month. Growth hormone measurements will occur on Day 23 after initiation of study drug administration
  Subjects will be given IM placebo/estradiol on Day 1. 10 days later they will receive IM placebo/estradiol again, then start progesterone/placebo capsules for 14 days. On Day 23, subjects will undergo a 12-h overnight (2200 - 1000h) fasting, 10-min blood sampling. A secondary outcome is GH secretion over the 2 hr after bolus ghrelin injection, a potent growth hormone secretagogue

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States